CLINICAL TRIAL: NCT01572363
Title: Fontan Patients: Comprehensive Evaluation of the Pulmonary Circulation to Identify Pulmonary Vascular Disease and Its Influence on Ventricular Hemodynamics.
Brief Title: Fontan Patients: Comprehensive Evaluation of Pulmonary Circulation and Ventricular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Alexander Van De Bruaene, Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ML6721
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Congenital Heart Disease
Keywords: Fontan; Cardiac magnetic resonance imaging; Sildenafil
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental): All patients will be given Sildenafil 50 mg with evaluation of pulmonary vascular resistance and systemic ventricular function at rest and during exercise after 30 minutes.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 50 mg once
  Other Names: Viagra; Revatio

SUMMARY:
In patients with one anatomical or functional ventricular chamber, which encompasses a spectrum of rare and complex congenital cardiac malformations, a staged surgical approach in view of an ultimate Fontan operation has become the procedure of choice. Especially in the earlier era, perioperative mortality was the leading cause of death. However, many patients have a long and high-quality life, continuously improved by a better understanding of Fontan hemodynamics and the refinement of the surgical procedures. Nevertheless, the prospect of eventual failure of the Fontan circulation remains a major concern. More specifically, evaluation of the pulmonary circulation becomes particularly important as the failing Fontan circulation has become a common indication for cardiac transplantation. Although essential, especially in the preoperative setting, a comprehensive evaluation of the pulmonary circulation remains difficult in this patient population

Our global hypothesis is that the absence of pulsatile pulmonary flow may lead to the development of pulmonary vascular lesions after the Fontan operation and that - together the absence of a subpulmonary ventricle for pressure generation - this increasing afterload will result in systemic ventricular underfilling and will eventually lead to a failing Fontan circulation.

DETAILED DESCRIPTION:
Background

In patients with one anatomical or functional ventricular chamber, which encompasses a spectrum of rare and complex congenital cardiac malformations, a staged surgical approach in view of an ultimate Fontan operation has become the procedure of choice. Especially in the earlier era, perioperative mortality was the leading cause of death. However, many patients have a long and high-quality life, continuously improved by a better understanding of Fontan hemodynamics and the refinement of the surgical procedures. Nevertheless, the prospect of eventual failure of the Fontan circulation remains a major concern. More specifically, evaluation of the pulmonary circulation becomes particularly important as the failing Fontan circulation has become a common indication for cardiac transplantation. Although essential, especially in the preoperative setting, a comprehensive evaluation of the pulmonary circulation remains difficult in this patient population.

Different types of Fontan circulation

Atriopulmonary connection

In the atriopulmonary connection, the right atrium is interposed as a valveless contractile chamber between the systemic venous and pulmonary arterial bed. Although initially believed to be beneficial, the interposition of such a valveless pulsatile chamber does not contribute positively to fluid energy. Moreover, pulsation results at the price of higher upstream pressures, whereas downstream pressures remain unchanged.

Total cavopulmonary shunts

This procedure consists of diverting the superior vena cava return into the pulmonary arteries and connecting the vena cava inferior to the pulmonary arteries. This action is achieved either by the construction of a composite conduit made of the sinus venarum and a prosthetic patch (intracardiac total cavopulmonary connection or lateral tunnel) or by an extracardiac conduit (extracardiac total cavopulmonary connection).

Our global hypothesis is that the absence of pulsatile pulmonary flow may lead to the development of pulmonary vascular lesions after the Fontan operation and that - together the absence of a subpulmonary ventricle for pressure generation - this increasing afterload will result in systemic ventricular underfilling and will eventually lead to a failing Fontan circulation.

Fontan attrition

The systemic ventricle

Although preload reduction may lead to inappropriate ventricular hypertrophy, with concomitant ventricular relaxation problems and a decreased capacity for adaptation to increased afterload, it is generally accepted that the pulmonary vasculature is more important than mild ventricular dysfunction in this patient population. Naturally, severe ventricular dysfunction will affect patient's prognosis.

The pulmonary circulation

The absence of a right ventricular to pulmonary arterial coupling has a profound influence on systemic venous return and the pulmonary circulation. Several aspects have to be taken into account when evaluating the pulmonary circulation

1. Systemic venous pressure.

   Systemic venous pressures, which are approximately 5 mmHg in healthy controls at rest and remains unchanged during exercise, are higher in Fontan patients. In Fontan patients, the absence of a right ventricle for pressure generation, some degree of congestion is required in order to force transpulmonary flow. However, at rest pressures above 20 mmHg are rarely seen as such pressures would lead to complications (oedema, pleural effusions and ascites). Interestingly, pressure change observed during exercise in normals and Fontan patients is quite similar. In healthy controls, an increase in mean pulmonary artery pressure from 15 mmHg at rest to 30 mmHg during exercise. In Fontan patients, mean right atrial pressure increased from 15 mmHg at rest to 25 mmHg during exercise.
2. Left atrial pressure.

   In healthy controls, left atrial pressures shows little variability at rest and is mainly determined by the atrioventricular valve and ventricular dysfunction. In Fontan patients, diastolic parameters are more difficult to assess as preload insufficiency should be considered.8 During exercise, left atrial pressure normally remains stable or increases somewhat in healthy individuals. However, there are few data available on left atrial pressures during exercise in Fontan patients.
3. Pulmonary circulation

Although there is still no unequivocal proof, several authors indicated that PVR appears to be the major determinant of cardiac output in Fontan patients at rest and during exercise. A low PVR is even more important in these patients as they do not have the possibility for adapting to a higher afterload, whereas in patients with a subpulmonary ventricle, increased afterload will be countered by RV hypertrophy. It has been suggested that Fontan patients having low PVR remain stable for many decades, whereas a high PVR appears to be poor prognostic factor.

Measurement of PVR and problems in Fontan patients

Most commonly, PVR is measured using the Fick method based on the principle that a known amount of a specific indicator is added to a volume of fluid. If the concentration before and after this addition is known, the volume of fluid can be calculated. The Fick method uses the physiological uptake of oxygen as an indicator. However, this method may be inaccurate in this patient population. Other techniques, such as the dye dilution technique or thermodilution technique suffer from their own limitations, such as reduced reliability in the presence of shunts or valvular regurgitation.

In order to provide a more accurate measurement of PVR, a combined approach of invasive pressure measurements and velocity-encoded magnetic resonance has become available, and has proven to be feasible in different patient populations. Cardiac output measured using this approach has been shown to be accurate and feasible in Fontan patients. Moreover, flow through to left and right pulmonary artery can be measured separately.

Measurement of PVR and ventricular volumes during exercise

As mentioned earlier, transpulmonary flow in Fontan patients is dependent on the presence of low PVR and normal behavior of PVR during exercise in order to be able to increase cardiac output. An increase in PVR during exercise would cause a more pronounced underfilling of the systemic ventricle with subsequently less increase or even decrease in stroke volume. Both pressure and flow measurements have been shown feasible in patients with congenital heart disease at rest and during exercise.

Measurement of PVR and ventricular volumes after vasodilatation Several studies have shown that drugs affecting the pulmonary vasculature (sildenafil, bosentan, NO) reduce PVR and increase cardiac output in selected patients. Especially in patients with elevated PVR, these drugs have the potential to decrease PVR and increase ventricular volumes, cardiac output and exercise tolerance. Whether these drugs improve outcome remains to be evaluated.

Aims of the study

Feasibility of measuring PVR in Fontan patients using simultaneous acquisition of invasive pressures and MR flow data.

Effect of Sildenafil 50 mg on PVR, ventricular volume and function at rest

Effect of bicycle stress on PVR, ventricular volume and function

Evaluating the reliability of bicycle stress echocardiography in determining ventricular volume and function as an indirect parameter reflecting the status of the pulmonary vasculature

ELIGIBILITY:
Inclusion Criteria:

* ≥ 14 years of age
* Written informed consent
* Fontan pathology

Exclusion Criteria:

* Inability to performe exercise
* Contra-indication for MR evaluation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Systemic ventricular stroke volume during exercise | 30 minutes after administration of sildenafil
  Systemic ventricular stroke volume during exercise as evaluated using bicycle stress magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium